CLINICAL TRIAL: NCT06288451
Title: DePTH: De-emphasize Parathyroid Hormone
Brief Title: DePTH: De-emphasize PTH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Simon Hsu, MD, MS, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00018021; 1K23DK136930-01 (NIH)
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are blinded to the assigned interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low dose oral calcitriol (Experimental)
  Interventions: Drug: Oral calcitriol with cinacalcet rescue
- Usual care (Active Comparator)
  Interventions: Drug: IV activated vitamin D

INTERVENTIONS:
Drug: Oral calcitriol with cinacalcet rescue — Participants will receive in-center oral calcitriol at a fixed dose of 0.5 mcg three times weekly at their dialysis treatment sessions regardless of their parathyroid hormone (PTH) concentrations over the 12-month trial period. Only if their serum PTH exceeds 800 pg/mL over 2 consecutive measurements will they be started on cinacalcet at 30 mg/d in order to protect against severe unremitting hyperparathyroidism.
  Arms: Low dose oral calcitriol
Drug: IV activated vitamin D — Participants will continue to receive intravenously-administered activated vitamin D per the Northwest Kidney Center treatment protocol, dose-titrated to monthly to quarterly parathyroid hormone concentrations.
  Arms: Usual care

SUMMARY:
The De-emphasize Parathyroid Hormone (DePTH) Study is a 12-month pragmatic, randomized, parallel-group, active comparator, open-label, blinded end-point study of 90 patients with incident or prevalent secondary hyperparathyroidism and kidney failure treated with in-center hemodialysis. It tests the hypothesis that low fixed-dose oral calcitriol (intervention) will have more favorable effects on a comprehensive panel of biomarkers that assesses mineral metabolism, bone turnover, and serum calcification propensity, compared with variably-dosed intravenous activated vitamin D titrated to PTH targets (usual care).

DETAILED DESCRIPTION:
Because of the kidneys' major role in vitamin D metabolism, most patients with kidney failure on dialysis have biochemical abnormalities that include vitamin D deficiency and high levels of phosphate, fibroblast growth factor-23 (FGF-23), and parathyroid hormone (PTH). All of these abnormalities are associated with cardiovascular disease, bone disease, and death and are major reasons why nephrologists have treated patients on dialysis with activated vitamin D agents for over 30 years. Current guidelines, however, encourage nephrologists to use high doses of vitamin D in order to lower PTH levels to pre-specified treatment targets. This approach to treatment has not been proven to improve health and survival, and may be associated with several harms, including further increasing levels of FGF-23 (a major cardiovascular risk factor), increasing calcium levels, which may promote vascular calcification, low turnover bone disease, and interruptions in vitamin D treatments.

Administering a low, stable dose of vitamin D may be safer and more effective than the current standard of care. The De-emphasize PTH (DePTH) Study is a pragmatic randomized clinical trial of 90 patients on hemodialysis in Seattle, WA, USA that tests whether a low fixed-dose of oral calcitriol (the active form of vitamin D; study intervention) is more safe, effective, and feasible compared with the current usual care. Participants will be recruited at their hemodialysis treatment centers and randomized in a 1:1 ratio to one of these two treatment strategies and followed over 12 months. Participants randomized to the study intervention will receive a fixed dose of calcitriol 0.5 mcg three times a week at their dialysis treatment sessions regardless of PTH level over the ensuing 12 months. Participants randomized to usual care will maintain the existing approach to treating abnormal mineral metabolism using vitamin D doses titrated to monthly to quarterly measurements of PTH. The outcomes for this trial are a panel of blood-based measurements of bone and vascular health that will be drawn at the same time as the blood work done monthly as part of routine dialysis care.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Kidney failure treated with in-center hemodialysis
3. PTH >=150 pg/mL x 2 consecutive measures at least 1 month apart or active IV activated vitamin D treatment using the NKC protocol

Exclusion Criteria:

1. History of parathyroidectomy or calciphylaxis
2. Severe secondary hyperparathyroidism (PTH >=600 pg/mL x 2 consecutive measures at least 1 month apart despite paricalcitol >=10 mcg 3x/week or doxercalciferol >=5 mcg 3x/week or cinacalcet >30 mg/d)
3. Calcium >9.8 mg/dL
4. Phosphate >9 mg/dL
5. Cholestyramine, phenytoin/phenobarbital, or ketoconazole use
6. Breast-feeding mothers
7. Inability to provide informed consent and no legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in fibroblast growth factor-23 | 12 months
  Change in fibroblast growth factor-23

SECONDARY OUTCOMES:
Change in serum calcium | 12 months
  Change in serum calcium
Change in serum phosphate | 12 months
  Change in serum phosphate
Change in serum bone-specific alkaline phosphatase | 12 months
  Change in serum bone-specific alkaline phosphatase
Change in serum parathyroid hormone | 12 months
  Change in serum parathyroid hormone
Change in T50 test of serum calcification propensity | 12 months
  Change in T50 test of serum calcification propensity

OTHER OUTCOMES:
Patient acceptability | 6 months
  Study acceptability to patients rated from 1 to 5 with 1 being the lowest acceptability and 5 being the highest
Patient acceptability | 12 months
  Study acceptability to patients rated from 1 to 5 with 1 being the lowest acceptability and 5 being the highest

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hsu, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No